CLINICAL TRIAL: NCT01160380
Title: A Phase III Study of Armodafinil for the Treatment of Cancer-Related Fatigue for Patients With Multiple Myeloma
Brief Title: A Study of the Effectiveness of Armodafinil to Treat Cancer-Related Fatigue in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: C10953/6270
Record Dates: First submitted 2010-07-07; First posted 2010-07-12 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Fatigue; Multiple Myeloma
Keywords: cancer related fatigue; fatigue; multiple myeloma; cancer; quality of life
MeSH Terms: conditions — Fatigue; Multiple Myeloma; Neoplasms | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armodafinil (Experimental): The patients receive armodafinil for all 56 days of the study.
  Interventions: Drug: armodafinil
- Placebo-First (Placebo Comparator): These patients receive a placebo for the first 28 days of the study. They are then crossed over and receive armodafinil for the final 28 days of the study (days 29-56).
  Interventions: Drug: armodafinil; Drug: Placebo

INTERVENTIONS:
Drug: armodafinil — Armodafinil taken at 150 mg daily. Taken as three 50 mg tablets.
  Other Names: Nuvigil
Drug: Placebo — Placebo taken at 150 mg daily. Taken orally as three 50 mg tablets.
  Other Names: sugar-pill
  Arms: Placebo-First

SUMMARY:
The purpose of this study is to evaluate the efficacy of armodafinil for the treatment of cancer-related fatigue in adult patients with multiple myeloma. The study consists of a screening period, followed by a 56-day treatment phase, and a final assessment to occur 28 days after the end of the last treatment.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, double-blind, randomized, placebo-controlled, crossover study to evaluate the efficacy of armodafinil at a dosage of 150 mg/day for the treatment of cancer-related fatigue (CRF) in adult patients with multiple myeloma. The study consists of a screening period, followed by a 56 day treatment phase, and a final assessment to occur 28 days after the end of the last treatment.

The screening period will occur within 14 days before baseline, where "baseline" refers to day 1 when assessments will be made before drug administration. During this period, a medical history will be obtained along with a complete physical examination including vital sign measurements and Eastern Cooperative Oncology Group (ECOG) performance status. Clinical laboratory tests including hematology, clinical chemistry (blood urea nitrogen [BUN], serum creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]), electrolytes (potassium, sodium, chloride and calcium), random glucose, total protein, albumin, and urinalysis will also be performed during the screening period as well as serum pregnancy tests for women of childbearing potential.

During the screening period, patients will also be assessed for the presence of cancer-related fatigue using the International Classification for Disease Tenth Edition (ICD-10) diagnostic criteria and the Brief Fatigue Inventory (BFI). Only those patients showing evidence of cancer-related fatigue will be enrolled in the study. The criteria for inclusion for any given patient consist of meeting the International Classification for Disease Tenth Edition (ICD-10) criteria for cancer-related fatigue and a score ≥ 4 on the BFI. ICD-10 CRF classification will be established using a standard interview guide.

Patients eligible for the study will be randomized to either receive armodafinil at an initial fixed dosage of 150 mg/day (Group A) or a placebo (Group B) during the first 28 days of the treatment phase. On day 29, patients randomized to receive placebo will then cross over to receive armodafinil at a dosage of 150 mg/day until day 56. Group A patients randomized to receive armodafinil will continue their current treatment with the drug until day 56. The duration of the treatment phase is 56 days.

Assessments for CRF will be conducted on day 1 (baseline) prior to drug treatment, and after drug administration on days 15, 28, 43, and 56. These assessments will be conducted as verbal interviews, paper-and-pencil surveys, paper-and-pencil tests, and electronic tests as appropriate per assessment.

During the treatment phase, each patient will also have clinical laboratory tests performed on days 1, 15, 28, 43 and 56 to monitor for potential toxicity. Additional procedures performed at these visits will include monitoring for adverse events, review of concomitant medications and other support therapies (e.g., growth factors and transfusion), ECOG performance status, vital signs measurements, and physical examinations.

Twenty-eight days after the last dose of study drug, patients are to complete a final assessment (herein referred to as the end-of-treatment visit). Procedures to be conducted at this visit include measurement of vital signs, a complete physical examination, assessment of adverse events, a review of concomitant medications, assessment of ECOG performance status, hematology and clinical chemistry laboratory tests including electrolytes, total protein and albumin. Patients who withdraw from the study before the completion of the 56 day cycle will still have all end-of-treatment assessments performed 28 days after their last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with multiple myeloma based on standard criteria
* The patient is diagnosed with cancer-related fatigue based on ICD-10 diagnostic criteria
* The patient shows signs of severe fatigue as evidenced by a Brief Fatigue Inventory score of at least 4
* The patient is a man or woman aged 18 years or older at the time of informed consent
* The patient has given voluntary written informed consent before any study-related procedure is performed which is not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Women of child bearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* Men must agree to use an acceptable method of contraception throughout the study and for 90 days after last dose study drug
* The patient must be willing and able to comply with study restrictions
* The patient must have an ECOG performance status not greater than 2
* The patient must have a life-expectancy of greater than 3 months
* The patient must meet the following laboratory criteria within 14 days of enrollment:

  * Platelet count greater than 50 x 109/L
  * Absolute neutrophil count greater than 0.5 x 109/L
  * Hemoglobin greater than 8 g/dL
  * AST and ALT not greater than 3.0 x the upper limit of normal (ULN)
  * Serum bilirubin not greater than 2.0 x ULN
  * Calculated or measured creatinine clearance of at least 10 mL/minute

Exclusion Criteria:

* The patient has been concurrently diagnosed with clinically significant depression
* The patient is concurrently enrolled in another investigational study that does not apply to the specific treatment of multiple myeloma
* The patient is receiving an investigational agent (non-FDA-approved) for any reason within 28 days of starting treatment on this study
* The patient has previously received armodafinil
* The patient has received modafinil or a psychostimulant within 14 days of enrollment
* The patient has received a blood transfusion within 14 days of enrollment
* The patient has impaired cardiac function or clinically significant cardiac diseases
* The patient has other concurrent severe and/or uncontrolled medical or psychiatric conditions including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* The patient has known positivity for human immunodeficiency virus (HIV) or hepatitis B or C; baseline testing for HIV and hepatitis B or C is not required
* The patient has undergone major surgery within 28 days of enrollment or has not recovered from side effects of such therapy (Kyphoplasty is not considered to be a major surgery; however, the investigator is to discuss enrollment of a patient with a recent history of kyphoplasty with Oncotherapeutics' medical monitor)
* The patient has a significant history of noncompliance to medical regimens or unwilling or unable to comply with the instructions given to him or her by the study staff
* The patient has a history of skin reactions and/or known sensitivity attributable to compounds of similar chemical or biological composition to modafinil, armodafinil, or the inactive ingredients in armodafinil including lactose monohydrate, starch, microcrystalline cellulose, croscarmellose, sodium, magnesium stearate or povidone
* The patient is a pregnant or lactating woman. Any women becoming pregnant during the study will be withdrawn from the study
* The patient is male whose sexual partner is a woman of childbearing potential not using effective birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, MD, Principal Investigator — James R. Berenson MD, Inc.
Locations (3):
- United States (3):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Michael J. Schlutz, M.D., Inc, Newport Beach, California
  - James R. Berenson, MD, Inc., West Hollywood, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Armodafinil: The patients receive armodafinil for all 56 days of the study.
  Armodafinil taken orally at 150 mg daily.
- Placebo-First: These patients receive a placebo for the first 28 days of the study. They are then crossed over and receive armodafinil for the final 28 days of the study (days 29-56).
  Placebo taken orally at 150 mg daily. Armodafinil taken orally at 150 mg daily.
Period: Overall Study
Arm/Group | Armodafinil | Placebo-First
Started | 25 | 25
Completed | 17 | 20
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Placebo-First | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (1.8) | 67 (2.3) | 65 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
ECOG (Eastern Cooperative Oncology Group) [Number; unit: paarticipants] — Grade ECOG Performance status
  0 Fully active, performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. Dead
  paarticipants
    0 | 5 | 7 | 12
    1 | 18 | 17 | 35
    2 | 2 | 1 | 3
Fatigue (baseline)-Brief Fatigue Inventory (BFI) [Median (Full Range); unit: units on a scale] — BFI scale: 9 items; range=0-90 (0-10 per item) Mild = 1-3 Moderate = 4-7 Severe = 8-10
  units on a scale | 59 [39 to 83] | 60.5 [36 to 79] | 60 [36 to 83]
Fatigue (baseline)-International Classification of Diseases version 10 (ICD-10) [Median (Full Range); unit: units on a scale] — ICD-10 Criteria (Range: 0-14) A1-A11 Fatigue Criteria B. Clinically significant distress or impaired functioning C. Symptoms are a consequence of cancer or cancer therapy D. Symptoms are a consequence of comorbid psychiatric disorders
  units on a scale | 9 [6 to 12] | 9 [6 to 12] | 9 [6 to 12]

OUTCOME MEASURES:

1. Primary Outcome: BFI Score
Description: Survey measuring fatigue. The scale contains 9 items; range=0-90 (0-10 per item). Mild = 1-3 Moderate = 4-7 Severe = 8-10
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
units on a scale
  Day 1(n=18, 23) | 65.0 (13.2) | 57.2 (14.3)
  Day 28 (n=19, 23) | 48.8 (22.4) | 41.5 (18.4)
  Day 56 (n=15) | 43.2 (18.9) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment; Test type: Superiority or Other; p = 0.289, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo-First; Comparison between Day 1 and Day 28; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Armodafinil; Comparison between Day 1 and day 28; Test type: Superiority or Other; p < 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Armodafinil; Comparison between Day 28 and Day 56 of treatment for the armodafinil arm; Test type: Superiority or Other; p = 0.449, t-test, 2 sided

2. Primary Outcome: Trail Making Test B Score (TMT-B)
Description: Cognitive test that gives a measure of various aspects of cognitive performance. Used to measure cognitive fatigue. The test consists of 25 circles containing 13 sequential numbers (1-13) and 12 sequential letters (A-L) positioned.
  The test evaluates the time to correctly order letters and numbers; low times = better performance.
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
seconds
  Day 1(n=18, 23) | 161.3 (77.8) | 220.5 (163.2)
  Day 28 (n=19, 23) | 158.4 (81.2) | 159.8 (94.2)
  Day 56 (n=15) | 153.8 (78.7) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment; Test type: Superiority or Other; p = 0.954, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Armodafinil; Day 1 vs. Day 28 of treatment for the Armodafinil arm; Test type: Superiority or Other; p = 0.369, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Armodafinil; Comparison between Day 28 and Day 56 of treatment for the Armodafinil arm; Test type: Superiority or Other; p = 0.973, t-test, 2 sided

3. Primary Outcome: Symbol Digit Modalities Test Score (SDMT)
Description: Test to evaluate neurocognitive functions (attention, visual scanning and motor speed). The test consists of a key =9 graphic symbols numbered 1 to 9 and the test =120 graphic symbols to be matched with its number. The test evaluates the number of correct matches within 90 seconds. Higher scores= better performance
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: Number of correct matches
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
Number of correct matches
  Day 1(n=18, 23) | 41.2 (9.2) | 40.7 (14.7)
  Day 28 (n=19, 23) | 42.4 (12.0) | 40.8 (14.7)
  Day 56 (n=15) | 48.7 (12.3) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms at day 28; Test type: Superiority or Other; p = 0.699, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm; Test type: Superiority or Other; p = 0.984, t-test, 2 sided
Statistical Analysis 3: Comparison: Armodafinil; Day 1 vs. Day 28 of treatment for the Armodafinil arm; Test type: Superiority or Other; p = 0.239, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Armodafinil; Day 28 vs. Day 56 of treatment for the Armodafinil arm; Test type: Superiority or Other; p = 0.089, t-test, 2 sided

4. Primary Outcome: Digit Span Test Score
Description: Test evaluates working memory and attention. The test consists of repeat numeric sequences of 2 to 9 numbers forward or backwards and evaluates the number of items from a sequence correctly named. Higher scores = better performance.
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: Number of correct items
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
Number of correct items
  Forward-Day 1 (n=18, 23) | 9.5 (2.7) | 9.8 (2.6)
  Backward-Day 1 (n=18, 23) | 7.3 (2.0) | 6.3 (2.4)
  Forward-Day 28 (n=19, 23) | 10.6 (3.0) | 10.4 (2.3)
  Backward- Day 28 (n=19, 23) | 7.0 (2.6) | 7.0 (2.6)
  Forward-Day 56 (n=15) | 10.3 (2.8) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  Backward-Day 56 (n=15) | 7.4 (2.8) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment for the Digit Span Test score-Forward test; Test type: Superiority or Other; p = 0.636, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment for the Digit Span Test score-Backward test; Test type: Superiority or Other; p = 0.531, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm-Digit Span Test score Forward test; Test type: Superiority or Other; p = 0.037, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm-Digit Span Test score Backward test; Test type: Superiority or Other; p = 0.656, t-test, 2 sided
Statistical Analysis 5: Comparison: Armodafinil; Day 1 vs. day 28 of treatment for the Armodafinil arm-Digit Span Test score-Forward test; Test type: Superiority or Other; p = 0.028, t-test, 2 sided
Statistical Analysis 6: Comparison: Armodafinil; Day 1 vs. day 28 of treatment for the Armodafinil arm-Digit Span Test score-Backward test; Test type: Superiority or Other; p = 0.805, t-test, 2 sided
Statistical Analysis 7: Comparison: Armodafinil; Day 28 vs. day 56 of treatment for the Armodafinil arm-Digit Span Test score-Forward test; Test type: Superiority or Other; p = 0.692, t-test, 2 sided
Statistical Analysis 8: Comparison: Armodafinil; Day 28 vs. day 56 of treatment for the Armodafinil arm-Digit Span Test score-Backward test; Test type: Superiority or Other; p = 0.863, t-test, 2 sided

5. Secondary Outcome: Functional Assessment of Cancer Therapy - Fatigue (FACIT-F) Score
Description: Survey addressing fatigue and patient happiness, coping, etc. Used to assess quality of life. The test consists of 40 items, each item with a response scale of 0-4. Higher scores denote better status Items are added to provide the total score (range 0-160).
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
units on a scale
  PWB-Day 1 (n=18, 23) | 14.1 (3.3) | 15.3 (5.1)
  SWB-Day 1 (n=18, 23) | 20.9 (6.7) | 19.8 (5.1)
  EWB-Day 1 (n=18, 23) | 16.9 (4.3) | 17.5 (3.7)
  FWB-Day 1 (n=18, 23) | 14.8 (3.6) | 14.6 (4.2)
  Fatigue-Day 1 (n=18, 23) | 19.2 (8.7) | 18.8 (8.9)
  FACIT-G-Day 1 (n=18, 23) | 67.0 (11.6) | 68.9 (11.4)
  TOI-Day 1 (n=18, 23) | 49.0 (12.2) | 49.4 (15.3)
  Total-Day 1 (n=19, 23) | 86.2 (15.8) | 86.1 (20.4)
  PWB-Day 28 (n=19, 23) | 16.5 (6.6) | 17.4 (6.3)
  EWB-Day 28 (n=19, 23) | 16.5 (5.3) | 18.7 (4.3)
  SWB-Day 28 (n=19, 23) | 21.3 (7.5) | 20.8 (5.4)
  FWB-Day 28 (n=19, 23) | 14.4 (5.1) | 16.8 (4.5)
  Fatigue-Day 28 (n=19, 23) | 28.0 (13.22) | 26.5 (11.7)
  FACIT-G-Day 28 (n=19, 23) | 68.5 (20.5) | 75.8 (12.9)
  TOI-Day 28 (n=19, 23) | 59.4 (23.5) | 62.9 (18.7)
  Total-Day 28 (n=19, 23) | 96.5 (31.3) | 101.3 (21.9)
  PWB-Day 56 (n=15) | 17.8 (5.1) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  EWB-Day 56 (n=15) | 22.1 (5.7) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  SWB-Day 56 (n=15) | 18.7 (3.4) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  FWB-Day 56 (n=15) | 13.5 (3.8) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  Fatigue-Day 56 (n=15) | 29.7 (9.2) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  FACIT-G-Day 56 (n=15) | 73.2 (12.1) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  TOI-Day 56 (n=15) | 62.7 (14.6) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  Total-Day 56 (n=15) | 101.8 (18.7) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms for Day 28 of treatment- FACIT-F total; Test type: Superiority or Other; p = 0.559, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm- FACIT-F total; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Armodafinil; Day 1 vs. Day 28 of treatment for the Armodafinil arm- FACIT-F total; Test type: Superiority or Other; p = 0.192, t-test, 2 sided
Statistical Analysis 4: Comparison: Armodafinil; Day 28 vs. Day 56of treatment for the Armodafinil arm- FACIT-F total; Test type: Superiority or Other; p = 0.495, t-test, 2 sided

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score
Description: Survey used to assess depression and anxiety. The test consists of 14 items (7 for anxiety and 7 for depression); there are 4 possible answers for each statement. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores= more anxiety or depression.
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
units on a scale
  Anxiety-Day 1 (n=18, 23) | 13.4 (21.4) | 8.3 (2.9)
  Depression-Day 1 (n=18, 23) | 7.8 (2.7) | 7.6 (3.2)
  Anxiety-Day 28 (n=19, 23) | 6.9 (4.6) | 5.5 (3.3)
  Depression-Day 28 (n=19, 23) | 10.3 (17.8) | 6.6 (3.6)
  Anxiety-Day 56 (n=15) | 7.0 (3.4) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
  Depression-Day 56 (n=15) | 5.7 (2.9) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment- HADS anxiety; Test type: Superiority or Other; p = 0.945, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Armodafinil vs Placebo-First; Comparison between arms at Day 28 of treatment- HADS depression; Test type: Superiority or Other; p = 0.316, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm-HADS anxiety; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm-HADS depression; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 5: Comparison: Armodafinil; Day 1 vs. Day 28 of treatment for the Armodafinil arm-HADS anxiety; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Armodafinil; Day 1 vs. Day 28 of treatment for the Placebo-First arm-HADS depression; Test type: Superiority or Other; p = 0.315, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Armodafinil; Day 28 vs. Day 56 of treatment for the Armodafinil arm-HADS anxiety; Test type: Superiority or Other; p = 0.933, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Armodafinil; Day 28 vs. Day 56 of treatment for the Armodafinil arm-HADS depression; Test type: Superiority or Other; p = 0.378, t-test, 2 sided

7. Secondary Outcome: Epworth Sleepiness Scale (ESS) Score
Description: Survey assessing sleep patterns. The test consists of 8 items. The response scale range is 0-24 (range 0-3 per item: 0-No chance to falling asleep; 3-high chance of falling asleep). Interpretation: 0-No chance to falling asleep; 10+ above average chance daytime sleepiness
Time Frame: Day 1, Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo-First
Number analyzed (Participants) | 25 | 25
units on a scale
  Day 1(n=18, 23) | 12.2 (5.1) | 11.5 (4.5)
  Day 28 (n=19, 23) | 10.1 (5.1) | 10.0 (4.6)
  Day 56 (n=15) | 11.5 (4.5) | NA (NA) — Day 56 data was only evaluated for the Armodafinil arm
Statistical Analysis 1: Comparison: Armodafinil vs Placebo-First; Comparison between arms for Day 28 of treatment -ESS; Test type: Superiority or Other; p = 0.840, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo-First; Day 1 vs. Day 28 of treatment for the Placebo-First arm-ESS; Test type: Superiority or Other; p = 0.050, t-test, 2 sided
Statistical Analysis 3: Comparison: Armodafinil; Day 1 and Day 28 of treatment for the Armodafinil arm- ESS; Test type: Superiority or Other; p = 0.051, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Armodafinil; Day 28 vs. Day 56 of treatment for the Armodafinil arm; Test type: Superiority or Other; p = 0.635, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Armodafinil: The patients receive armodafinil for all 56 days of the study.
  Armodafinil taken orally at 150 mg daily. All patients receiving armodafinil, including patients that crossover, were evaluated for adverse events (AEs) and serious adverse events (SAEs).
- Placebo-First: These patients receive a placebo for the first 28 days of the study. They are then crossed over and receive armodafinil for the final 28 days of the study (days 29-56).
  Placebo taken orally at 150 mg daily. Armodafinil taken orally at 150 mg daily.
  AEs presented were those occurring during from Day 1 to Day 28 only
Arm/Group | Armodafinil | Placebo-First
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/25
Other Adverse Events (participants affected / at risk) | 15/50 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=50) | Placebo-First (N=25)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ptosis (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (N=50) | Placebo-First (N=25)
G3/G4 Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
G3/G4 Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
G3/G4 Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
G3/G4 BUN (increased) (Renal and urinary disorders) | 1 (1) | 0 (0)
G3/G4 Creatinine (increased) (Renal and urinary disorders) | 1 (1) | 0 (0)
G4 Edema (General disorders) | 1 (1) | 0 (0)
G3/G4 Eosinophils (increased) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
G3/G4 Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
G3/G4 Infection (ear) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
G3/G4 Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
G3/G4 Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No